CLINICAL TRIAL: NCT04927325
Title: Quantification of Erythema at Exit Site of Central Catheter: Is a Tablet Camera Sufficient?
Brief Title: Erythema at Exit Site & Tablet Camera
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christina Hafner, Clinical Investigator, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1165/2021
Record Dates: First submitted 2021-06-02; First posted 2021-06-16 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2021-12

CONDITIONS: CLABSI - Central Line Associated Bloodstream Infection; CRBSI - Catheter Related Bloodstream Infection; Digital Technology

STUDY DESIGN:
Intervention Model Description: 10 central lines with a reddened exit site 10 central lines without a reddened exit site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- central line with a reddened exit site (Other): A standardized set of photos will be taken of 10 central lines with an erythema at exit site (visible to the naked eye)
  Interventions: Other: Set of Photos
- Control Group: central line without a reddened exit site (Other): A standardized set of photos will be taken of 10 newly inserted CVC (as a control over time to evaluate the in-patient redness and the impact of irritation of a CVC)
  Interventions: Other: Set of Photos

INTERVENTIONS:
Other: Set of Photos — A standardized set of photos will be taken with a tablet camera, SLR, thermal camera.

SUMMARY:
Background: In critical care medicine central venous catheters play an important role in the source of infections. In the daily routine prior to the diagnosis the suspicion of catheter related infection is discussed in the medical team due to signs of systemic inflammation or exit site infection like erythema, induration or tenderness. However, if an erythema at exit site of a central line can be quantified with a tablet camera, is unknown.

Methods: Standardized set of photos will be taken of 10 central lines with a reddened exit site and 10 catheters without an erythema (as a control over time) with a tablet camera and a single-lens reflex camera. The percentage of usable images between tablet and single-lens reflex camera will be analysed. Furthermore, two independent clinical experts from dermatology will grade blinded de-identied images on a scale from 0 to 4 (0 - no erythema, 1- very faint, 2 - faint, 3 - bright, 4 - very bright).

Objectives: The primary objective of this feasibility study aims to analyze the reliability of a tablet camera as a device for quantification of erythema around an exit site.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Jugular CVC or Subclavian CVC
* ICU-Admission

Exclusion Criteria:

* < 18 years
* Pregnancy/Lactation
* HIV
* neutropenia (<1000/m3)
* hematologic tumor
* dark pigmentation
* prone position within the last 24 hours
* head/neck-area: cancer, operation, burns or radiation, tattoos

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Percentage of usable images | through study completion, an average of 3 months
  The percentage of useable images of tablet camera compared with single-lens reflex (SLR) camera will be analysed.

SECONDARY OUTCOMES:
Quantification of the exit site with regards to an erythema scale | through study completion, an average of 3 months
  The secondary objective aims to evaluate the quantification of the exit site regarding to the erythema scale by two independent clinical experts comparing images of tablet and SLR camera.
  The erythema will be graded using a visual ordinal scale (grade 0 to grade 4). Grade 0 represents no erythema, whereas grade 4 describes a very bright erythema.

CONTACTS AND LOCATIONS:
Overall Officials: Department of Anaesthesia & General Intensive Care, Study Chair — Medical University of Vienna
Locations (1):
- Department of Anesthesia, General Intensive Care and Pain Management,Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No